CLINICAL TRIAL: NCT01642459
Title: The Outcomes of Arteriovenous Fistula (AVF) Cannulated From Different Direction in Maintenance Hemodialysis Patients.
Brief Title: The Outcomes of Arteriovenous Fistula Cannulated From Different Direction.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The patients enrolled are limited.
Sponsor: Dongliang Zhang, MD (Other)
Responsible Party: Sponsor-Investigator, Dongliang Zhang, MD, Associated professer, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-0107
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Arteriovenous Fistula
Keywords: arteriovenous fistula; hemodialysis; aneurysm; vascular stenosis; cannulation
MeSH Terms: conditions — Arteriovenous Fistula; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Same direction cannulation (Experimental): The inserted direction of arterial needle is same as the direction of blood flow.
  Interventions: Other: Same direction cannulation
- Opposite direction cannulation (Active Comparator): The inserted direction of arterial needle is opposite to the direction of blood flow.
  Interventions: Other: Opposite direction cannulation

INTERVENTIONS:
Other: Same direction cannulation — The puncture direction of the arterial needle is same as the blood flow in every hemodialysis session.
  Arms: Same direction cannulation
Other: Opposite direction cannulation — The puncture direction of the arterial needle is opposite to the blood flow in every hemodialysis session.
  Arms: Opposite direction cannulation

SUMMARY:
The investigators hypothesis that aneurysms and stenoses will be decreased if the direction of inserted arterial needle were same as the direction of blood flow, when compared to the opposite direction puncture.

DETAILED DESCRIPTION:
Native arteriovenous fistula (AVF) is the preferred access for hemodialysis, and cannulation technique is very important factors affect the outcomes of AVF. Rope-ladder cannulation is one kind of the standard puncture techniques which is used commonly in maintenance hemodialysis (MHD) patients. There are many complications for rope-ladder cannulation, such as venous aneurysm and vascular stenosis, which may induce AVF dysfunction. For the venous outflow way, there always be aneurysm followed by stenoses at the sites of needle connected with the arterial line in rope-ladder cannulation patients. The investigators hypothesis that the directions of inserted arterial needles should affect the AVF outcomes. The present prospective study will compare the outcomes of AVF between the puncture direction at arterial needle sites same as blood flow and opposite to blood flow.

ELIGIBILITY:
Inclusion Criteria:

* MHD patients with autogenous AVF.
* Newly setup AVF in 3 months.
* Fore- or Upper arm AVF.
* Flow of >800ml/min detected by using the ultrasound dilution technique.

Exclusion Criteria:

* AVF after neoplasty.
* Arteriovenous grafts.
* Anticipated live time less than one year.
* Patients whose concurrent illnesses, disability, or geographical residence would hamper attendance at required study visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of AVF aneurysm and stenosis. | 12 months
  Compare the prevalence of AVF aneurysm and stenosis between two groups during 12 months.

SECONDARY OUTCOMES:
Proportions of AVF dysfunction in different groups. | 12 months
  Compare the proportions of AVF dysfunction between two groups during 12 months.
The size of venous aneurysm. | 12 months
  Measure the maximum size of venous aneurysm by using ultrasonography at month 12.
Diameter of venous stenosis. | 12 months
  Measure the minimum diameter of venous stenosis by ultrasonography at month 12.
Percentages of unsuccessful cannulations. | 12 months
  Unsuccessful cannulations include mis-cannulation, cannulation ease, hematoma, more than once cannulation at arterial site.
Events of AVF obstruction. | 12 months
  AVF obstruction and the following treatments as central venous catheters and interventions will be recorded and compared between two groups during 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dongliang Zhang, Doctor, Study Chair — Kidney Disease Faculty of Capital Medical University; Wenying Cui, Bachelor, Study Director — Nephrology Department of Beijing Friendship Hospital
Locations (1):
- Beijing Friedship Hospital, Beijing, Beijing Municipality, China